CLINICAL TRIAL: NCT01625871
Title: Artemether/Lumefantrine in the Treatment of Plasmodium Vivax Malaria in Eastern Sudan
Brief Title: Artemether/Lumefantrine and Vivax Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Khartoum (Other)
Collaborators: University of Kassala, Sudan (Other)
Responsible Party: Principal Investigator, Ishag Adam, Professor, University of Khartoum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: vivax
Record Dates: First submitted 2012-06-17; First posted 2012-06-22 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Vivax Malaria
Keywords: malaria; vivax; artemether/lumefantrine; Sudan
MeSH Terms: conditions — Malaria, Vivax; Malaria | interventions — Artemether; Lumefantrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- artemether-lumefantrine (Experimental): tablets (containing 20mg artemether and 120 mg lumefantrine) for three days
  Interventions: Drug: tablets artemether/lumefantrine

INTERVENTIONS:
Drug: tablets artemether/lumefantrine — six doses of oral tablets of artemether/lumefantrine
  Other Names: Quartem

SUMMARY:
The cure rate of artemether/lumefantrine in the treatment of vivax malaria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vivax malaria

Exclusion Criteria:

* severe malaria
* pregnancy

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The cure rate | 28 days
  The proportion of the cure patients

SECONDARY OUTCOMES:
Fever clearance time | 28 days
  The time for fever clearance
Parasite clearance time | 28 days
  The time for the parasite to clear

CONTACTS AND LOCATIONS:
Locations (1):
- Kassala, Kassala, Kassala, Sudan

REFERENCES:
- [Background] Makanga M, Krudsood S. The clinical efficacy of artemether/lumefantrine (Coartem). Malar J. 2009 Oct 12;8 Suppl 1(Suppl 1):S5. doi: 10.1186/1475-2875-8-S1-S5. PMID 19818172
- [Derived] Abdallah TM, Ali AA, Bakri M, Gasim GI, Musa IR, Adam I. Efficacy of artemether-lumefantrine as a treatment for uncomplicated Plasmodium vivax malaria in eastern Sudan. Malar J. 2012 Dec 5;11:404. doi: 10.1186/1475-2875-11-404. PMID 23217037
- See also: http://www.ncbi.nlm.nih.gov/pubmed?term=adam%20i — http://www.ncbi.nlm.nih.gov/pubmed?term=adam%20i